CLINICAL TRIAL: NCT03855605
Title: Evaluation of Algorithm for Diagnosis of Hypertension by Home Blood Pressure Monitoring
Brief Title: Diagnosis of Hypertension by Home Blood Pressure Monitoring
Status: Completed | Type: Observational
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Moo-Yong Rhee, Professor, Principal Investigator, DongGuk University
Other Study IDs: DUMC-C1502
Record Dates: First submitted 2019-02-24; First posted 2019-02-27 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Hypertension,Essential; Home Blood Pressure; Ambulatory Blood Pressure
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Home blood pressure measurement has been recommended to use in the diagnosis of hypertension. The investigators have developed diagnostic algorithm of hypertension by using 24-hour and home blood pressure measurement. However, the diagnostic agreement between home blood pressure measurement and 24-hour ambulatory blood pressure measurement is about 70 - 85%. The discrepancy of diagnosis between home blood pressure measurement and 24-hour ambulatory blood pressure is one of the barriers to introduce home blood pressure measurement in the diagnosis of hypertension.

To solve the discrepancy, identifying the characteristic patients showing discrepancy of hypertension diagnosis between home blood pressure measurement and 24-hour ambulatory blood pressure measurement is needed.

The purpose of the present study are (1) to validate the diagnostic algorithm of hypertension by using 24-hour ambulatory blood pressure and home blood pressure measurement the investigators have developed, and (2) to identifying the characteristics of patients showing discrepancy of diagnosis between 24-hour ambulatory blood pressure and home blood pressure measurement, and (3) lastly to improve the diagnostic algorithm of hypertension by using home blood pressure measurement.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Patients with high blood pressure measured by doctors at the outpatient office

Exclusion Criteria:

* Patients taking antihypertensive drugs or blood pressure affecting drugs within 1 month
* Secondary hypertension
* Hypertensive emergency and urgency
* Severe heart failure (NYHA III and IV)
* Angina with 6 months
* Myocardial infarction within 6 months
* Peripheral artery disease within 6 months
* Significant arrhythmia (i.e. ventricular tachycardia and fibrillation, atrial fibrillation, atrial flutter)
* Pregnancy
* Night labor, shift worker
* Those who are currently participating in other clinical studies
* Those who have taken other clinical trial drugs within the past month
* According to the opinion of the researcher, those who have or may have a disease that may interfere with the completion of the study
* History of drug or alcohol dependence within 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At the out-patient clinics, study investigators recruit study participants who have high blood pressure measured by them at the out-patient clinics and adequate for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
validation of the diagnostic algorithm of hypertension | at baseline
  validation of the diagnostic algorithm of hypertension by using 24-hour ambulatory blood pressure and home blood pressure measurement

SECONDARY OUTCOMES:
the characteristics of patients showing discrepancy of diagnosis | at baseline
  the characteristics of patients showing discrepancy of diagnosis between 24-hour ambulatory blood pressure and home blood pressure measurement
the change of diagnostic discrepancy | from baseline to more than 6 months
  the change of diagnostic discrepancy between 24-hour ambulatory blood pressure and home blood pressure measurement during follow up period more than 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
In order to share the individual participant data, the informed consent from the research participants is required un the Korean law, and we did not get the consent to share at the beginning of this study.

REFERENCES:
- [Derived] Lee YJ, Rhee MY, Kim JS, Do U, Kim JH, Kim BK, Kim HY. Association of the magnitude of the difference in blood pressure between office and ambulatory measurements with blood pressure variability in untreated individuals. Clin Hypertens. 2022 Dec 15;28(1):36. doi: 10.1186/s40885-022-00220-7. PMID 36517899